CLINICAL TRIAL: NCT06117501
Title: Nerve Protection Evaluation: Revision Cubital Tunnel Syndrome Decompression
Acronym: COVERED
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Axogen Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANP-CP-001
Record Dates: First submitted 2023-10-27; First posted 2023-11-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Cubital Tunnel Syndrome; Recalcitrant Cubital Tunnel Syndrome
Keywords: Cubital Tunnel Syndrome; Revision Cubital Tunnel Surgery; First Revision Cubital Tunnel Syndrome Decompression; Ulnar Nerve; Ulnar Nerve Neuropathy; Nerve Protection; Axoguard HA+ Nerve Protector
MeSH Terms: conditions — Cubital Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- First Revision Cubital Tunnel with application of Axoguard HA+ Nerve Protector (Other): Single group assignment. Patients will receive the Axoguard HA+ Nerve Protector™ in their first revision cubital tunnel surgery.
  Interventions: Device: Axoguard HA+ Nerve Protector™

INTERVENTIONS:
Device: Axoguard HA+ Nerve Protector™ — Axoguard HA+ Nerve Protector™ is a surgical implant that provides non-constricting protection for non-transected peripheral nerve injuries where there is no gap. Axoguard HA+ Nerve Protector™ is designed to be an interface between the nerve and the surrounding tissue.

SUMMARY:
This single-cohort, prospective case series is designed to evaluate and characterize the use of Axoguard HA+ Nerve Protector™ to protect the ulnar nerve in a first revision cubital tunnel decompression procedure. Data on the primary cubital tunnel syndrome decompression, first revision decompression utilizing Axoguard HA+ Nerve Protector, participant-reported pain, motor and sensory functional outcomes, quality of life (QoL) outcomes, and recurrence/revision will be collected. This case series will help to establish the ability of Axoguard HA+ Nerve Protector to provide clinical benefits for patients undergoing a first revision cubital tunnel decompression procedure.

DETAILED DESCRIPTION:
The objectives of this study are:

1. To evaluate the use and characterize the performance of Axoguard HA+ Nerve Protector to protect the ulnar nerve in a first revision cubital tunnel decompression by understanding post-operative outcomes (pain level, QoL, PROMs, and ulnar nerve specific functional outcomes) compared to baseline (pre-revision operative levels).
2. To summarize the safety of Axoguard HA+ Nerve Protector, an FDA-cleared device, in first revision cubital tunnel decompression procedures.
3. To characterize the feasibility of Axoguard HA+ Nerve Protector to prevent the recurrence of compressive neuropathy of the ulnar nerve at the elbow and resulting need for future revision procedures.
4. To characterize the feasibility of imaging the ulnar nerve pre- and post-operatively to assess nerve and tissue bed health.

The study population includes participants 18 years of age or older presenting for evaluation of surgery for compressive ulnar nerve neuropathy at the elbow following a primary cubital tunnel syndrome decompression.

Data will be collected from available medical records and patient reported outcomes questionnaires using approved data collection forms (paper or electronic). The following data will be collected at the respective study visits: demographics, primary decompression details, revision decompression details, baseline assessments, health-related QoL questionnaires, functional assessments, and recovery assessments.

There will be a total of nine (9) study visits (Pre-op Screening/Baseline and Operative Day visits plus seven (7) study follow-up events).

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 18 years of age;
2. Have symptoms of ulnar nerve neuropathy near the elbow present at 180 days or greater following a primary cubital tunnel decompression procedure.
3. Be eligible for surgical intervention;
4. Have a preoperative diagnostic such as a nerve conduction study, electromyography, or ultrasound evaluation documenting ulnar neuropathy at the elbow;
5. Have a baseline pain visual analogue scale (VAS) score due to ulnar nerve neuropathy of no less than 40/100 mm for the affected elbow;
6. Have at least one of the following:

   * Paresthesia or numbness in the ulnar nerve distribution;
   * Weakness or wasting of the small muscles of the hand (full hand muscle wasting is excluded);
   * A positive elbow flexion provocation test.
7. Undergo a first revision cubital tunnel decompression surgery with placement of Axoguard HA+ Nerve Protector circumferentially around the section of ulnar nerve affected by neuropathy;
8. Be willing and able to comply with all aspects of the treatment and evaluation schedule over 18 months; and
9. Sign and date an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved written informed consent prior to initiation of any study procedures.

Exclusion Criteria:

1. Have had a previous revision cubital tunnel decompression procedure;
2. Have documented evidence of concomitant neuropathic conditions affecting the subject arm or any proximal condition affecting the subject arm including, but not limited to:

   * Previously treated carpal tunnel syndrome with unresolved symptoms or current carpal tunnel syndrome that will not be treated concurrently with the revision cubital tunnel;
   * Cervical or brachial plexus abnormalities or injuries;
   * Cervical spine or shoulder disease;
   * Thoracic outlet syndrome;
   * Complex regional pain syndrome;
   * Polyneuropathy, systemic neuropathy or Lyme disease related neuropathy;
   * Previous or current surgery of the ulnar nerve at the wrist (Guyon's canal release)
   * Ulnar nerve compression at the wrist/Guyon's canal;
3. Have current trauma or past trauma with ongoing pathology that interferes with evaluation or treatment of the ulnar nerve to either side shoulder or upper extremity;
4. Have previous radiofrequency ablation, presence of nerve stimulator or received nerve implant(s) in the subject arm or be receiving an implant(s) other than Axoguard HA+ Nerve Protector during the study surgical procedure, that will impact the ulnar nerve or planned study evaluations;
5. Have a condition(s) that could confound assessments or health-related quality of life including, but not limited to:

   * Rheumatoid arthritis
   * Fibromyalgia
   * Connective tissue disorder
   * Wrist tenosynovitis
6. Be a smoker or tobacco user;
7. Currently have or have a history of alcohol or drug abuse;
8. Have uncontrolled Diabetes Mellitus at the discretion of the treating surgeon or have diabetic neuropathy in the upper extremities;
9. Have documented poorly controlled hyperthyroidism or hypothyroidism;
10. Have a known sensitivity to porcine derived materials or those containing hyaluronate or alginate or their components;
11. Be currently taking or likely to need medication(s) that may cause or contribute to peripheral neuropathy or peripheral nerve dysfunction at the discretion of the treating surgeon;
12. Be taking prescribed medication(s) including, but not limited to, narcotics 2 or more times per week for the treatment of chronic pain or chronic nerve related symptoms NOT associated with the subject ulnar nerve neuropathy; or
13. Be deemed unsuitable for inclusion in the study at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 6-18 months
  Change from baseline in visual analog scale (VAS) pain scores (0-100 mm) will be evaluated between post-operative months 6 to 18 to characterize treatment response over time.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 3 months
  Pain will be assessed on each study visit using a 100 mm visual analog scale (VAS).
Grip strength | 18 months
  Grip strength will be measured for both arms using a hand dynamometer.
Semmes-Weinstein Monofilament test | 18 months
  Semmes-Weinstein Monofilament test will be performed to assess sensibility by evaluating the tactile sensitivity to pressure in both hands to pressure applied by the monofilaments.
Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) score | 18 months
  QuickDASH is a patient-reported outcome questionnaire to measure physical functions and symptoms in patients with upper limb musculoskeletal disorders including cubital tunnel syndrome. The QuickDASH is scored in two components: the disability/symptom section (11 items, scored 1-5) and the optional high performance sport/music or work modules (four items, scored 1-5).
Patient-Reported Outcomes Measurement Information System® (PROMIS®) Bank v2.1 Upper Extremity | 18 months
  PROMIS® is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. The PROMIS Bank v2.1 - Upper Extremity is a patient questionnaire developed to assess upper extremity physical function in patients with hand and upper extremity conditions as a separate domain from general physical function.
Patient-Rated Ulnar Nerve Evaluation (PRUNE) | 18 months
  The Patient-Rated Ulnar Nerve Evaluation (PRUNE) score is a brief, open-access, patient-reported outcome measure specifically for patients with ulnar nerve compression at the elbow that assesses pain, symptoms and functional disability.
Modified McGowan classification | 18 months
  McGowan classification grades the severity of CuTS based on patient-reported symptoms and physical examination findings.
12-Item Short Form Health Survey (SF-12) | 18 months
  The 12-Item Short Form Health Survey (SF-12) is a self-reported, health-related quality of life questionnaire assessing the impact of health on an individual's everyday life.

OTHER OUTCOMES:
Proportion of participants with healthy ulnar nerve appearance | 18 months
  Sponsor-developed qualitative questionnaire assessing nerve health by imaging the nerve using ultrasound or MRI. Scale describes nerve as healthy (normal) or unhealthy (abnormal) in appearance.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Foundation for Orthopaedic Research and Education (Florida Orthopaedic Institute), Tampa, Florida
  - Optim Orthopedics, Savannah, Georgia
  - Indiana Hand to Shoulder Center, Indianapolis, Indiana
  - University of New Mexico, Albuquerque, New Mexico
  - Cleveland Clinic, Cleveland, Ohio
  - Rothman Orthopaedics, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No